CLINICAL TRIAL: NCT07290686
Title: Evaluation of the Effectiveness and Safety of an Innovative, Non-pharmacological Method Using Transcranial Direct Current Stimulation in Combination With Cognitive Training and Nasal Near Infrared Stimulation to Improve Cognitive Functions and Quality of Life in Elderly People With Mild Cognitive Impairment (MCI) and Alzheimer's Disease (AD).
Brief Title: Evaluation of the Effectiveness and Safety of Transcranial Direct Current Stimulation in Combination With Nasal Near Infrared Stimulation to Improve Cognitive Functions and Quality of Life in Elderly People With Mild Cognitive Impairment (MCI) and Alzheimer's Disease (AD).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Jakub Kazmierski, MD PhD Professor of Medical University of Lodz, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RNN/336/20/KE
Record Dates: First submitted 2023-12-14; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Active tDCS stimulation (Active Comparator): 50 sessions of active stimulation of current intensity 2mA, stimulation time 20 minutes
  Interventions: Device: tDCS stimulation
- Placebo tDCS stimulation (Placebo Comparator): 50 sessions of sham stimulation lasting only 30 seconds
  Interventions: Device: tDCS
- Active iNIRS stimulation (Active Comparator): 50 sessions of active stimulation of intranasal near- infrared of 850 wavelength IR diode
  Interventions: Device: iNIRS stimulation
- Placebo iNIRS stimulation (Placebo Comparator): 50 sessions of sham stimulation lasting only 30 seconds
  Interventions: Device: iNIRS

INTERVENTIONS:
Device: tDCS stimulation — tDCS delivered with the anode at F3 (according to the 10-20 EEG electrode mounting system) and the cathode in F4, covering the left and right dorsolateral frontal cortexes, respectively.
  Arms: Active tDCS stimulation
Device: tDCS — tDCS delivered with the anode at F3 (according to the 10-20 EEG electrode mounting system) and the cathode in F4, covering the left and right dorsolateral frontal cortexes, respectively.
  Arms: Placebo tDCS stimulation
Device: iNIRS stimulation — intra-nasal
  Arms: Active iNIRS stimulation
Device: iNIRS — intra-nasal
  Arms: Placebo iNIRS stimulation

SUMMARY:
Alzheimer's disease (AD) and mild cognitive impairment (MCI) are progressive neurodegenerative conditions with limited therapeutic options. Today, around 30 million people worldwide suffer from Alzheimer's dementia. According to WHO predictions, the number of people affected by Alzheimer's disease in 2030 will amount to 65 million, and in 2050 nearly 115 million This means that the number of people suffering from Alzheimer's disease will triple in the next 30 years. The exact cause of Alzheimer's disease is still unknown. The amyloid hypothesis assumes that the accumulation of insoluble β-amyloid 42 aggregates in the central nervous system (CNS) triggers tau hyperphosphorylation (taupathy) and neurodegeneration in AD from the preclinical stage to dementia. In the 1990s, pharmacological treatment of Alzheimer's disease was introduced, but numerous studies indicate its limited effectiveness. Despite many attempts, there is currently no effective drug to delay the course of Alzheimer's disease. In recent years, there have been scientific reports indicating that the use of neuromodulatory therapies has a positive effect on the cognitive functions, behavior and daily functioning of AD patients.

Neuromodulation techniques such as transcranial direct current stimulation (tDCS) and photobiomodulation (PBM) have shown promise in improving cognitive function, but their combined effects remain underexplored.

The aim of the current project is to develop an effective and safe therapeutic procedure based on transcranial direct current stimulation (tDCS) therapy enriched with near infrared nasal stimulation (iNIRS) in patients diagnosed with mild cognitive impairment (MCI) and Alzheimer's disease (AD).

DETAILED DESCRIPTION:
The aim of the current project is to develop an effective and safe therapeutic procedure based on transcranial direct current stimulation (tDCS) therapy enriched with cognitive training and near infrared nasal stimulation (iNIRS) in patients diagnosed with mild cognitive impairment (MCI) and Alzheimer's disease (AD) . The project will also evaluate the effectiveness of the selected therapeutic method and its impact on the improvement of cognitive functions of patients, including memory, attention, concentration, executive and language functions, as well as the presence of neuropsychiatric symptoms / behavioral disorders in patients and the quality of life of patients.

People meeting the inclusion criteria will be invited to participate in the study and will be provided with and written information about the research project and a voluntary, informed consent form.

Clinical evaluation of patients using the following scales: Mini Mental State Examinaton, Alzheimers Disease Assessment Scale, Neuropsychiatric Inventory Questionnaire, Geriatric Depression Scale, Hachiński Ischemic Index, Rey-RAVLT Fifteen Words Test. Cognitive assessments were performed at baseline, at the end of the procedure (within the three days after the last treatment session), and after 12 weeks of follow-up.

Clinical and demographic data: age, sex, education, the course of the disease to date, comorbidities, medications taken, smoking.

Patients will be randomly assigned to two parallel research groups - an active group receiving combination therapy with tDCS with cognitive exercise and nasal near infrared stimulation and placebo group with tDCS sham without cognitive training and sham nasal stimulation.

The procedure will include daily (5 out of 7 days a week) tDCS sessions lasting a total of 20 minutes. tDCS will be delivered at 2 mA with the anode at F3 (according to the 10-20 EEG electrode mounting system) and the cathode in F4, covering the left and right dorsolateral frontal cortexes, respectively.

During the tDCS procedure, patients received intranasal near-infrared stimulation through the device, utilizing an IR diode with the following parameters: 850nm wavelength, 40Hz pulse frequency, and a 50% duty cycle. Stimulation was administered for 20 minutes, five days a week, consecutively. Both stimulations were administered simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MCI/AD
* MMSE 12-26 points
* ADAS- COG > 17 points
* signed inform consent form
* minimum 8 years of education
* stable drug doses for minimum 3 months

Exclusion Criteria:

* diagnosis of mental disability, schizophrenia, bipolar disorder, depression, alcohol and/or drug addiction,
* unstable somatic state
* lack of signed inform consent form

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
cognitive functions assessed by MMSE scale | up to 12 weeks
  change over time of cognitive functions measured as a change in amount of points during MMSE scale assestment. Change will be evaluated as overall reasult of scale and also as result in every assest field (according to MMSE scale). Assessment conducted on baseline, up to 3 days after end of the procedure and after 12 weeks.
cognitive functions assessed by ADAS- Cog scale | up to 12 weeks
  change over time of cognitive functions measured as a change in amount of points during ADAS-Cog scale assestment. Change will be evaluated as overall reasult of scale and also as result in every assest field (according to ADAS-Cog scale). Assessment conducted on baseline, up to 3 days after end of the procedure and after 12 weeks.
cognitive functions assessed by RAVLT | up to 12 weeks
  change over time of cognitive functions measured as a change in amount of points during RAVLT assestment. Change will be evaluated as overall reasult of scale and also as result in every assest field (according to RAVLT). Assessment conducted on baseline, up to 3 days after end of the procedure and after 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Old Age Psychiatry and Psychotic Disorders Medical University of Lodz, Lodz, Łódź Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No